CLINICAL TRIAL: NCT04989049
Title: Main Objective While Treating the Ulcers is to Reduce the Discomfort and Accelerate Healing. Thus the Purpose of the Study is to Find Out Therapeutic Role of Topical Folic Acid on Oral Ulcerations
Brief Title: Therapeutic Effect of Folic Acid in Healing of Oral Ulcers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tahseen Shabbir Khooharo, post graduate trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: folic acid for oral ulcers
Record Dates: First submitted 2021-07-07; First posted 2021-08-04 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Oral Ulcer
Keywords: folic acid; oral ulcers; topical therapy
MeSH Terms: conditions — Oral Ulcer | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: 75 patients divided into two groups 35 in each
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group or case group (Active Comparator): topical folic acid on oral ulcers will be applied for 7 days and patients will be asked to visit after 7 days for follow up
  Interventions: Drug: Folic Acid 5 MG
- control group (Placebo Comparator): placebo drug for oral ulcers
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Folic Acid 5 MG — folic acid tablet of 5mg will be placed on the ulcers 2 times per day for 7 days
  Other Names: folacin
  Arms: intervention group or case group
Other: placebo — an inactive drug looking exactly like active drug will be given, patients will be asked to put it on ulcers 2 times per day
  Other Names: inactive drug
  Arms: control group

SUMMARY:
patients reporting at the department of oral medicine with the complain of oral ulceration will be asked to participate in this study.

DETAILED DESCRIPTION:
Oral ulcerations are usually reported with pain and discomfort while eating and drinking at times while talking. Ulcers are usually described as erythematous surroundings, raised margins, with yellowish-white necrotic pseudomembranous centre. Healing process of ulcers usually starts nearly after 24-48 h of its onset. The initial inflammatory stage is enriched by leukocytes, after 48 hours of injury, mature monocytes in connective tissue turn into macrophages which until day 3 tend to increase in numbers. Oral ulcers are one of the commonest lesions of oral cavity; around 83.6% people have suffered from the ulcers. Frequency of traumatic ulcers fluctuates from 3 to 34% around the globe. Traumatic ulcers are usually caused by mechanical irritaation. Various studies have been conducted till date for the treatment of oral ulcers such as anti-inflammatory gels, propolis extract gel, topical steroids such as triamcinolone acetonide paste and silver nanoparticle gel.

Folic acid (vitamin b9) belongs to the water soluble class of vitamins called B-complex. It is an essential component of metabolic pathways of carbohydrates, fats and proteins which are important compounds in various functions such as cardiovascular and nervous system. This vitamin is also important for DNA methylation and biosynthesis of nucleotide. Dietary foliate deficiency is a problem of developing country. Folic acid daily requirement of an adult is 400 mg/day whereas during pregnancy it's required up to 600mg and in nursing mother daily required dosage of foliate is 500mg/day.

The difference between folic acid and foliate is that the foliate is a natural form which is found in mushrooms, green leafy vegetables and livers whereas folic acid is synthetically produced and is used to fortify processed foods and supplements in a fully reduced biologically active form dihydrofolate reductase. Humans lack the enzyme which is required to produce foliate that is why they depend on dietary and supplemental form of this essential vitamin.

Main objective while treating the ulcers is to reduce the discomfort and accelerate healing. Thus the purpose of the study is to find out therapeutic role of topical folic acid on oral ulcerations.

Patients falling in the inclusion criteria will be asked to participate in the study, consent will be obtained from the patients. Demographic feature, history and examination will be noted on a research questionnaire. After examination patients will be given topical folic acid in tablet form to be applied by themselves twice a day on ulcers. Patients will be asked to visit the dental out patients department of oral medicine at Isra University Hyderabad on 7th day for follow up. Specific questions will be asked from the patients and examination will be done on the day of follow, the information will be recorded on a follow up form.

ELIGIBILITY:
Inclusion Criteria:

* • Age of the participant will be between 14 to 44 years old

  * Both of the genders will be included
  * Patients with oral ulceration

Exclusion Criteria:

* • Reluctant to participate

  * Non healing ulcerations, lasting for more than 14 days after removing the cause
  * Patients with neurological problems, psoriasis, rheumatoid arthritis.

Ages: 14 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
healing of ulcers | 7 days
  patients will be examined to evaluate if the ulcers are healed completely, follow up questionnaire form will be filled by the examining dentist, describing the condition of the patient.

IPD SHARING:
Plan to Share IPD: No